CLINICAL TRIAL: NCT05101057
Title: A Retrospective Study to Examine the Effect of Adjuvant Combined Magnetic Field Stimulation on Primary Anterior Cervical Discectomy and Fusion (ACDF) Patients
Brief Title: A Retrospective Study to Examine the Effect of CMF Stimulation on Primary ACDF Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-608
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-10

CONDITIONS: Degeneration of Cervical Intervertebral Disc

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Treated: Patients who underwent ACDF surgery and who received post surgical therapy with the SpinalogicTM Non-Invasive Bone Graft Stimulation Device.
  Interventions: Device: SpinalogicTM Bone Graft Stimulator
- Control: Patients who underwent ACDF surgery and did not receive post surgical Bone Graft Stimulation.

INTERVENTIONS:
Device: SpinalogicTM Bone Graft Stimulator — The SpinalogicTM is a portable, battery-powered, microprocessor-controlled, non-invasive bone growth stimulator. The device is currently approved and commercially indicated as an adjunct electrical treatment to primary lumbar spinal fusion surgery for one or two levels.
  Groups: Treated

SUMMARY:
A retrospective parallel group comparison study to support expansion of the indication of the company's FDA approved Spinalogic™ device to include the cervical spine. The SpinalogicTM device was initially approved by FDA as an adjunct to one- or two-level lumbar fusion (P910066/S011). It is a non-invasive bone growth stimulator (BGS) that generates a combined magnetic field (CMF) that has been proven to accelerate bone healing and fusion in the lumbar spine.

ELIGIBILITY:
Inclusion Criteria

* Male or Female aged 18-75 years.
* Primary anterior cervical discectomy fusion (ACDF) and required two level spinal fusion or were active smokers and required either single or two level spinal fusion.
* Pain VAS score >5 and/or extreme weakness at target operative level(s).
* At least one post operative clinical outcome assessment (VAS pain/ NDI/OC score) at each follow up interval.
* Completed 6 month follow up visit or time to fusion assessment, whichever is sooner.

Exclusion Criteria

* Treated with a bone growth stimulator device other than the SpinalogicTM CMF device.
* Previous cervical vertebrae fusion surgery at any level (posterior or anterior approach)
* Systemic administration of any type of corticosteroid, antineoplastic, immune- stimulating or immunosuppressive agents within 30 days of primary ACDF surgery and/or within 12 weeks post-operatively.
* Active history of systemic malignancy at pre-operative assessment or during 12- month follow up period.
* Untreated malignant neoplasm(s) or underwent radiotherapy or chemotherapy at pre- operative assessment or during 12-month follow up period.
* Implanted with cardiac pacemaker or implantable cardioverter defibrillator at pre- operative assessment or during 12-month follow up period.
* Pregnant at pre-operative assessment or during 12-month follow up period.
* Mental or physical condition that would interfere with post-treatment assessments and/or care (e.g., neuromuscular disease, psychiatric disease,
* Paraplegia, quadriplegia, etc.) at pre-operative assessment or during 12-month follow up period.
* Prescribed non-steroidal anti-inflammatory, calcium channel blockers and/or diphosphonate therapy within 12-weeks of surgery period.
* Prescribed bone morphogenic protein (BMP) during 12-month follow up period.
* Implanted with a Titanium cage during the primary ACDF that precludes an outcome determination via plain radiographs.
* Osseous or ligamentous spinal trauma at pre-operative assessment or during 12- month follow up period.
* Paget's disease at pre-operative assessment or during 12-month follow up period.
* Absence of X-ray fusion assessment documentation at 6 months follow-up visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects underwent primary anterior cervical discectomy and fusion (ACDF) and required two- level cervical spine fusions. OR were active smokers and required either single or two-level cervical spine fusions.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to fusion | 12 months
  Comparison of the cervical fusion rate between treated and control group patients

SECONDARY OUTCOMES:
Patient Reported Outcome Measures VAS | 12 months
  VAS Pain Score
Patient Reported Outcome Measures NDI | 12 months
  Neck Disability Index
Patient Reported Outcome Measures OC | 12 months
  Odum's Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ruba Sarris, MPH, Study Director — DJO
Locations (2):
- United States (2):
  - SIOSD, San Diego, California
  - BSSNY, White Plains, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez-Lara A, Nandyala SV, Fineberg SJ, Singh K. Current trends in demographics, practice, and in-hospital outcomes in cervical spine surgery: a national database analysis between 2002 and 2011. Spine (Phila Pa 1976). 2014 Mar 15;39(6):476-81. doi: 10.1097/BRS.0000000000000165. PMID 24365907
- [Background] Eck JC, Hodges SD, Humphreys SC. Techniques for stimulating spinal fusion: efficacy of electricity, ultrasound, and biologic factors in achieving fusion. Am J Orthop (Belle Mead NJ). 2001 Jul;30(7):535-41. PMID 11482508
- [Background] Gruskay JA, Webb ML, Grauer JN. Methods of evaluating lumbar and cervical fusion. Spine J. 2014 Mar 1;14(3):531-9. doi: 10.1016/j.spinee.2013.07.459. Epub 2013 Oct 31. PMID 24183750
- [Background] Veeravagu A, Cole T, Jiang B, Ratliff JK. Revision rates and complication incidence in single- and multilevel anterior cervical discectomy and fusion procedures: an administrative database study. Spine J. 2014 Jul 1;14(7):1125-31. doi: 10.1016/j.spinee.2013.07.474. Epub 2013 Oct 11. PMID 24126076
- [Background] Leven D, Cho SK. Pseudarthrosis of the Cervical Spine: Risk Factors, Diagnosis and Management. Asian Spine J. 2016 Aug;10(4):776-86. doi: 10.4184/asj.2016.10.4.776. Epub 2016 Aug 16. PMID 27559462
- [Background] Hilibrand AS, Fye MA, Emery SE, Palumbo MA, Bohlman HH. Impact of smoking on the outcome of anterior cervical arthrodesis with interbody or strut-grafting. J Bone Joint Surg Am. 2001 May;83(5):668-73. doi: 10.2106/00004623-200105000-00004. PMID 11379735
- [Background] Campbell PG, Yadla S, Nasser R, Malone J, Maltenfort MG, Ratliff JK. Patient comorbidity score predicting the incidence of perioperative complications: assessing the impact of comorbidities on complications in spine surgery. J Neurosurg Spine. 2012 Jan;16(1):37-43. doi: 10.3171/2011.9.SPINE11283. Epub 2011 Oct 28. PMID 22035101